CLINICAL TRIAL: NCT06998914
Title: Arthroscopic Assisted Distal Radius Fracture Fixation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Mansour Mohamed, residant doctor, Assiut University
Other Study IDs: Arthro distal radius fix
Record Dates: First submitted 2025-04-14; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Radius Fracture
MeSH Terms: conditions — Radius Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Recent distal radius fractures which occurred less than 14 day clssification 2R3B1,2R3B2,2R3B3,2R3C1 on AO classification with articular surface displacement or gap ≥ 2mm after reduction

SUMMARY:
Distal radius fractures (DRF) are among the most common orthopedic injuries, both in young adults and in elderly patients.(1,2,4،7 ) Effective management of these fractures is crucial to restoring wrist function, ensuring stability, and minimizing complications. (2)Traditional open reduction and internal fixation (ORIF) remains the cornerstone of treatment. (3)However, minimally invasive techniques are increasingly gaining attention for their ability to improve outcomes while reducing complications.(5, 8) Wrist arthroscopy has emerged as a valuable tool in the management of DRF. It allows for direct visualization of intra-articular fractures, assessment of associated soft tissue injuries, and precise reduction of fracture fragments. Additionally, it facilitates the identification and management of concomitant injuries, such as triangular fibrocartilage complex (TFCC) tears or ligament injuries, which are frequently overlooked in traditional techniques. (6, 9 ،10) Despite these advantages, the use of wrist arthroscopy in DRF management remains underutilized in many regions. In Assiut University Hospital, there is a growing interest in incorporating advanced techniques, including wrist arthroscopy, into the management of orthopedic injuries. However, there is limited local data on the outcomes and feasibility of this approach in the treatment of DRF. This case series aims to evaluate the clinical and functional outcomes of DRF management using wrist arthroscopy, providing insight into its effectiveness, safety, and applicability in a tertiary care setting. By documenting the experiences and outcomes of patients treated with this innovative technique, this study seeks to contribute to the existing literature and guide the future adoption of arthroscopy-assisted methods in DRF management in the region.

-The aim of this study is to evaluate the clinical and functional outcomes of managing distal radius fractures assisted by wrist arthroscopy at Assiut University Hospital using Mayo wrist score, with a focus on its effectiveness, safety, and feasibility in improving fracture reduction, identifying associated injuries, and enhancing patient recovery.

ELIGIBILITY:
Inclusion Criteria:

* Recent distal radius fractures which occurred less than 14 day clssification 2R3B1,2R3B2,2R3B3,2R3C1 on AO classification with articular surface displacement or gap ≥ 2mm after reduction
* Patient aged from 18 to 60 years.
* Potential associated ligament injuries.

Exclusion Criteria:

* Poly-traumatized patients or those with other fractures in the same upper limb.
* Open fractures or neurovascular deficit or medical fractures.
* Patient with severe complications that prevent clear visualization during arthroscopy.
* Patient with uncontrolled chronic diseases, especially uncontrolled DM or HTN

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Recent distal radius fractures which occurred less than 14 day clssification 2R3B1,2R3B2,2R3B3,2R3C1 on AO classification with articular surface displacement or gap ≥ 2mm after reduction
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
healing of radius fracture | 6 month
  evaluate distal radius fracture treated by wrist arthroscopy using The X-ray beam was centered 1 m above the radius fracture. Anteroposterior (AP) and lateral films (LAT) were taken Four orthopedic surgeons with similar ranks were chosen and blindly asked to evaluate three parameters of radiographic measurements for each set of radiographs.